CLINICAL TRIAL: NCT00350727
Title: Phase I and II, Open-Label, Multi-Center Trials of Pazopanib in Combination With Lapatinib in Adult Patients With Relapsed Malignant Glioma
Brief Title: Pazopanib In Combination With Lapatinib In Adult Patients With Relapsed Malignant Glioma
Acronym: VEG102857
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG102857; NCT00412711 (obsolete NCT alias)
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Results first posted 2011-06-20 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2012-05

CONDITIONS: Glioma
Keywords: relapsed; lapatinib; Pazopanib; glioblastoma
MeSH Terms: conditions — Glioma; Recurrence; Glioblastoma | interventions — pazopanib; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination (Experimental): Pazopanib and Lapatinib in combination. Subjects remain on treatment until disease progression or withdrawal from study.
  Interventions: Drug: pazopanib; Drug: lapatinib

INTERVENTIONS:
Drug: pazopanib — Pazopanib is a novel compound being developed for the treatment of various cancers.
Drug: lapatinib — Lapatinib is a novel compound being developed for the treatment of various cancers.
  Other Names: pazopanib

SUMMARY:
This study is being conducted to characterize the safety/tolerability of pazopanib and lapatinib when administered in combination with enzyme-inducing anticonvulsants in patients with recurrent Grade III or IV malignant gliomas.

DETAILED DESCRIPTION:
This study is being conducted to characterize the safety/tolerability of pazopanib and lapatinib when administered in combination with enzyme-inducing anticonvulsants in patients with recurrent Grade III or IV malignant gliomas.

ELIGIBILITY:
Inclusion criteria:

Phase I

* Patients are on EIAC for a minimum of 15 days. Patients may be on more than one anti-convulsant (AC). At least one of the ACs must be an EIAC.
* Patients with anaplastic astrocytoma, anaplastic oligodendroglioma, mixed anaplastic oligoastrocytoma, glioblastoma multiforme, or gliosarcoma at recurrence
* Patients whose diagnostic pathology confirmed these pathologies will not need re-biopsy
* Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to Grade III or IV malignant glioma Phase II
* Patients must have histologically confirmed glioblastoma multiforme or gliosarcoma in first or second recurrence.
* Patients may not have received more than two prior cytotoxic chemotherapy containing regimen.
* Patients must not have received prior treatment with VEGFR, ErbB1, ErbB2 inhibitors including but not limited to PTK-787, Sorafenib, Sutent, Tarceva, Iressa, Erbitux, and Herceptin. Prior Avastin therapy is permitted provided three months has elapsed before Day 1, Treatment Period 1.
* Tumor tissue must be analyzed for PTEN and epidermal growth factor receptor (EGFR) vIII prior to dosing.
* Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to Grade IV malignant glioma.
* Patients must not be on an EIAC. NOTE: Once the (optimally tolerated regimen) OTR in Phase I is determined and all patients in the expanded cohort have completed 1 treatment period then patients on EIAC may be enrolled in the Phase II component of the study.

Phase I and II

* Male or female, age at least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) status 0 to 1 as per protocol.
* Clinical lab results as per protocol
* Has a left ventricular ejection fraction (LVEF) at least 50% based on echocardiogram (ECHO) or Multi Gated Aquisition (MUGA) or within the institutional normal range.
* Adequate renal function
* Creatinine clearance more than 50 mL/min as calculated by the Cockcroft-Gault formula as per protocol.
* Urine Protein Creatinine (UPC) ratio of less than or equal to 1 as per protocol.
* Able to swallow and retain oral medications.
* A woman is eligible to enter and participate in the study if she is of:

  - Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:
* Has had a hysterectomy,
* Has had a bilateral oophorectomy (ovariectomy),
* Has had a bilateral tubal ligation,
* Is post-menopausal (total cessation of menses for at least 1 year)

  - Childbearing potential, has a negative serum pregnancy test at screening, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female patient's entry and is the sole sexual partner for that female.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
* A man with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.
* If sexually active, patients will continue the recommended contraceptive measures for the duration of the treatments and for 28 days following discontinuation of therapy.
* Signed informed consent approved by the Institutional Review Board prior to patient entry.

Exclusion criteria:

* Poorly controlled hypertension as per protocol. NOTE: Initiation or adjustment of BP medication is permitted prior to study entry provided that patient has two consecutive BP readings less than 140/90 mmHg each separated by a minimum of 24 hrs. These readings need to be collected prior to enrolment.
* Concurrent severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive cardiac failure, poorly controlled hypertension, history of labile hypertension, history of poor compliance with antihypertensive regimen, chronic renal disease, or active uncontrolled infection) that could compromise participation in the study.
* History of myocardial infarction, admission for unstable angina, cardiac angioplasty or stenting within three months of Day 1, Treatment Period 1.
* Has Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system as per protocol.
* QTc prolongation defined as a corrected QT (QTc) interval greater than or equal to 470 milliseconds.
* History of venous or arterial thrombosis within 3 months of Day 1, Treatment Period 1.
* Current use of therapeutic warfarin. NOTE: both low molecular weight heparin and prophylactic low-dose warfarin are permitted; however, prothrombin time/partial thromboplastin time (PT/PTT) must meet above inclusion criteria.
* Excessive risk of bleeding as defined by stroke within the prior 6 months, history of central nervous system (CNS) or intraocular bleed, or septic endocarditis.
* Evidence of intratumor hemorrhage on pretreatment diagnostic imaging, except for stable post-operative Grade 1 hemorrhage.
* Active systemic bleeding, such as gastrointestinal bleeding or gross hematuria.
* Female patients who are pregnant or breast feeding.
* Acute or chronic liver disease (i.e., hepatitis, cirrhosis).
* Patients who received investigational drugs less than 21days prior to Day 1, Treatment Period 1, or who have not recovered from the toxic effects of such therapy.
* Patients who received chemotherapy less than or equal to 21days prior (6 weeks for prior nitrosourea or mitomycin C) to Day 1, Treatment Period 1, or who have not recovered from the toxic effects of such therapy.
* Patients who received radiation therapy less than or equal to 12 weeks prior to Day 1, Treatment Period 1, or who have not recovered from the toxic effects of such therapy as per protocol.
* Patients who received biologic, immunotherapeutic or cytostatic agents less than or equal to 14 days prior to Day 1, Treatment Period 1, or who have not recovered from the toxic effects of such therapy.
* Patient is less than 3 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant or requiring active intervention. Patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Surgical resection of brain tumor or any other surgery less than or equal to 21 days prior to Day 1, Treatment Period 1, or who have not recovered from side effects of such a procedure. Patients who undergo stereotactic biopsy less than or equal to 14 days prior to Day 1 of Treatment Period 1, or who have not recovered from side effects of such a procedure.
* Patients with any Grade of intraparenchymal CNS hemorrhage. Exceptions include Grade 1 intraparenchymal hemorrhage in the immediate post-operative period, or Grade 1 intraparenchymal hemorrhage that has been stable for at least 3 months.
* Patients unwilling to or unable to comply with the protocol.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with patient safety or obtaining informed consent.
* History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism or excretion of study drugs. Has any unresolved bowel obstruction or diarrhea.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Is on any specifically prohibited medication or requires any of these medications during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] de Jonge MJ, Hamberg P, Verweij J, Savage S, Suttle AB, Hodge J, Arumugham T, Pandite LN, Hurwitz HI. Phase I and pharmacokinetic study of pazopanib and lapatinib combination therapy in patients with advanced solid tumors. Invest New Drugs. 2013 Jun;31(3):751-9. doi: 10.1007/s10637-012-9885-8. Epub 2012 Oct 6. PMID 23054212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I and Phase II had two separate participant populations. Enrollment in Phase II was not dependent on the number of participants completing Phase I.
Groups:
- Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg: Starting dose of oral pazopanib of 200 milligrams (mg) once daily (OD) and oral lapatinib 1500 mg OD. The dose of pazopanib (200-800 mg) and lapatinib (500-1500 mg) in cohorts enrolled subsequent to the first dose cohort was determined by the toxicity profile of the combination therapy and the pharmacokinetic results from the prior cohort.
- Phase II: Biomarker Positive: All participants received pazopanib 400 mg twice daily (BID) and lapatinib 1000 mg OD. Biomarker-positive participants were those who expressed epithelial growth factor receptor vIII (EGFRvIII) and/or phosphate and tensin homolog (PTEN).
- Phase II: Biomarker Negative: All participants received pazopanib 400 mg OD and lapatinib 1000 mg OD. Biomarker-negative participants were those who did not express either EGFRvIII and/or PTEN.
Period: Phase I: Dose Escalation
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Started | 34 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 34 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Lack of Efficacy | 25 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Transition to Extension Phase | 3 | 0 | 0
Period: Phase II
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Started | 0 | 19 | 22
Completed | 0 | 0 | 0
Not Completed | 0 | 19 | 22
Not completed — Disease Progression | 0 | 15 | 16
Not completed — Clinical Deterioration | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Death | 0 | 0 | 2
Not completed — Sponsor Terminated Study | 0 | 0 | 1
Not completed — Enrolled in Rollover Study | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative | Total
Number analyzed (Participants) | 34 | 19 | 22 | 75
Age, Customized [Number; unit: participants] — Number of participants falling into the indicated age groups.
  participants
    20-29 years old | 1 | 0 | 2 | 3
    30-39 years old | 8 | 0 | 3 | 11
    40-49 years old | 11 | 6 | 6 | 23
    50-59 years old | 10 | 5 | 8 | 23
    60-69 years old | 3 | 7 | 2 | 12
    >=70 years old | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 5 | 21
  Male | 23 | 14 | 17 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 0 | 0 | 1 | 1
  White/Caucasian/European Heritage | 34 | 19 | 21 | 74

OUTCOME MEASURES:

1. Secondary Outcome: Phase I: Pharmacokinetic Parameters Including AUC(0-24), [AUC(0-12) for Patients on Twice Daily Administration], Cmax, the Time to Maximum Observed Concentration (Tmax) and C24 of Pazopanib and Lapatinib When Administered in Combination With EIAC.
Time Frame: Completed during first cycle of treatment.
Reporting Status: Not Posted

2. Secondary Outcome: Phase II: Pharmacokinetic Parameters Including AUC(0-24), [AUC(0-12) for Patients on Twice Daily Administration], Cmax, Tmax, and C24 of Pazopanib and Lapatinib, as Appropriate, When Administered Together in Combination With Non-EIAC.
Time Frame: Completed during first cycle of treatment.
Reporting Status: Not Posted

3. Secondary Outcome: Phase II: Plasma Concentrations of the Circulating Biomarkers VEGF, sVEGFR-1, and sVEGFR-2.
Time Frame: Completed during first cycle of treatment.
Reporting Status: Not Posted

4. Primary Outcome: Number of Participants With the Indicated Change From Baseline to Study Completion in Systolic Blood Pressure
Description: Each on-study and follow-up laboratory parameter and vital sign was compared to the participant's baseline (BL) values to investigate what changes occurred. mmHg, millimeters of mercury.
Time Frame: Baseline to study completion (up to 844 days for Phase I, up to 878 days for Phase II)
Population: All-treated Population (all participants who were given any dose of study medication) for Phases I and II. One participant withdrew in Phase I due to death; change from baseline was not calculated for this participant.
Measure: Number; unit: participants
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 33 | 19 | 22
participants
  BL, 90-<140 mmHg; shift to post-BL, 90-<140 mmgHg | 21 | 12 | 11
  BL, 90-<140 mmHg; shift to post-BL, 140-<170 mmHg | 12 | 3 | 8
  BL, 90-<140 mmHg; shift to post-BL, >=170 mmHg | 0 | 0 | 1
  BL, 140-<170 mmHg; shift to post-BL, 90-<140 mmHg | 0 | 1 | 0
  BL, 140-<170 mmHg; shift to post-BL, 140-<170 mmHg | 0 | 2 | 1
  BL, 140-<170 mmHg; shift to post-BL, >=170 mmHg | 0 | 0 | 0
  BL, >=170 mmHg; shift to post-BL, 140-<170 mmHg | 0 | 1 | 1

5. Primary Outcome: Number of Participants With the Indicated Change From Baseline to Study Completion in Diastolic Blood Pressure
Description: as for outcome 4
Time Frame: Baseline to study completion (up to 844 days for Phase I, up to 878 days for Phase II)
Population: All-treated Population for Phases I and II. One participant withdrew in Phase I due to death; change from baseline was not calculated for this participant.
Measure: Number; unit: participants
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 33 | 19 | 22
participants
  BL, 50-<90 mmHg; shift to post-BL, 50-<90 mmHg | 23 | 13 | 9
  BL, 50-<90 mmHg; shift to post-BL, 90-<110 mmHg | 9 | 4 | 10
  BL, 90-<110 mmHg; shift to post-BL, 50-<90 mmHg | 0 | 1 | 0
  BL, 90-<110 mmHg; shift to post-BL, 90-<110 mmHg | 1 | 0 | 2
  BL, 90-<110 mmHg; shift to post-BL, >=110 mmHg | 0 | 1 | 1

6. Primary Outcome: Number of Participants With the Indicated Change From Baseline to Study Completion in Heart Rate
Description: Each on-study and follow-up laboratory parameter and vital sign was compared to the participant's baseline (BL) values to investigate what changes occurred. bpm, beats per minute.
Time Frame: Baseline to study completion (up to 844 days for Phase I, up to 878 days for Phase II)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 33 | 19 | 22
participants
  BL, 44-100 bpm; shift to post-BL, 44-100 bpm | 31 | 14 | 19
  BL, 44-100 bpm; shift to post-BL, 101-120 bpm | 0 | 3 | 2
  BL, 101-120 bpm; shift to post-BL, 101-120 bpm | 2 | 0 | 0
  BL, 101-120 bpm; shift to post-BL, >120 bpm | 0 | 1 | 0
  BL, >120 bpm; shift to post-BL, 44-100 bpm | 0 | 0 | 1
  BL, missing; shift to post-BL, 44-100 bpm | 0 | 1 | 0

7. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Albumin
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: All-treated Population for Phase II. Data are presented for only those participants who provided chemistry measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 21
grams per liter (g/L) | -5.9 (9.57) | -6.7 (9.95)

8. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, and Lactate Dehydrogenase
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
International Units per Liter (IU/L)
  Alkaline phosphatase, n=19, 21 | 18.6 (54.02) | 33.9 (109.99)
  Alanine aminotransferase, n=19, 22 | 56.1 (131.99) | 132.7 (393.89)
  Aspartate aminotransferase, n=19, 22 | 36.4 (88.50) | 52.7 (178.02)
  Lactate dehydrogenase, n=18, 19 | 291.50 (443.725) | 171.63 (606.986)

9. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Amylase and Lipase
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 19
Units per liter (U/L)
  Amylase | 22.72 (28.060) | 20.05 (30.288)
  Lipase | 131.4 (318.13) | 120.5 (163.51)

10. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Total Bilirubin and Creatinine
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/l)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 21
micromoles per liter (µmol/l)
  Total bilirubin | 6.174 (7.2714) | 23.562 (71.1671)
  Creatinine | 6.93 (10.444) | 9.59 (14.852)

11. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Calcium, Glucose, Potassium, Magnesium, Inorganic Phosphorus, Sodium, and Urea
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/l)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 21
millimoles per liter (mmol/l)
  Calcium, n=19, 21 | 0.004 (0.1257) | 0.019 (0.0952)
  Glucose, n=19, 21 | 0.082 (4.1342) | 1.850 (2.7180)
  Potassium, n=19, 21 | 0.17 (0.471) | 0.30 (0.264)
  Magnesium, n=19, 19 | 0.022 (0.0676) | 0.040 (0.0853)
  Sodium, n=19, 21 | 1.7 (2.96) | 1.3 (1.85)
  Urea, n=19, 21 | 0.770 (1.6840) | 1.071 (2.1736)
  Inorganic phosphorus, n=19, 20 | 0.090 (0.2352) | 0.076 (0.2048)

12. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Thyroxine and Free T3 (Triiodothyronine)
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/l)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 16 | 13
picomoles per liter (pmol/l)
  Thyroxine, n=16, 13 | -8.052 (30.2175) | 10.806 (40.5626)
  Free T3, n=4, 4 | 0.420 (0.5010) | -2.442 (2.3525)

13. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Thyroid Stimulating Hormone
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliunits per liter (mU/L)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 18 | 20
milliunits per liter (mU/L) | 1.37 (2.106) | 2.59 (4.377)

14. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Total T3
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/l)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 13 | 8
nanomoles per liter (nmol/l) | -0.181 (0.6521) | -0.104 (0.3516)

15. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Hemoglobin
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: All-treated Population for Phase II. Data are presented for only those participants who provided hematology measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
grams per liter (g/L) | -4.6 (11.25) | -8.0 (16.75)

16. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Hematocrit
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline. The hematocrit is the proportion of blood volume that is occupied by red blood cells.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
percent | -0.016 (0.0320) | -0.027 (0.0452)

17. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Lymphocytes, Neutrophils, Platelet Count, and White Blood Count
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: giga (10^9) per liter (GI/L)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
giga (10^9) per liter (GI/L)
  Lymphocytes, n=16, 19 | -0.26 (0.556) | -0.21 (0.573)
  Total Neutrophils, n=16, 18 | -2.87 (3.021) | -4.72 (5.067)
  Platelet count, n=19, 22 | -58.7 (53.98) | -55.7 (59.79)
  White blood cells, n=19, 22 | -2.63 (2.934) | -4.06 (6.026)

18. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for International Normalized Ratio (Prothrombin Time)
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline. Prothrombin time is a measure of the extrinsic pathway of coagulation that is used to determine the clotting tendency of blood. The International Normalized Ratio is the ratio of a patient's prothrombin time to a normal (control) sample.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: All-treated Population for Phase. Data are presented for only those participants who provided hematology measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
ratio | 0.030 (0.0663) | 0.042 (0.1094)

19. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase II of the Study for Partial Thromboplastin Time and Prothrombin Time
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline. Partial thromboplastin time is a performance indicator detecting abnormalities in blood clotting.
Time Frame: Baseline to study completion (up to 878 days for Phase II)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
seconds (sec)
  Partial thromboplastin time | 2.10 (1.985) | 2.62 (3.175)
  Prothrombin time | 0.0 (0.57) | 0.2 (1.19)

20. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Albumin
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: All-treated Population for Phase I. Data are presented for only those participants who provided chemistry measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Groups:
- Phase I: Pazopanib 200 mg /Lapatinib 1500 mg: Pazopanib 200 mg OD and Lapatinib 1500 mg OD
- Phase I: Pazopanib 800 mg /Lapatinib 1500 mg: Pazopanib 800 mg OD and Lapatinib 1500 mg OD
- Phase I: Pazopanib 800 mg/Lapatinib 500 mg: Pazopanib 800 mg OD and Lapatinib 500 mg BID
- Phase I: Pazopanib 800 mg/Lapatinib 750 mg: Pazopanib 800 mg OD and Lapatinib 750 mg BID
- Phase I: Pazopanib 800 mg/Lapatinib 1000 mg: Pazopanib 800 mg OD and Lapatinib 1000 mg BID
- Phase I: Pazopanib 600 mg/Lapatinib 1000 mg: Pazopanib 600 mg BID and Lapatinib 1000 mg BID
Arm/Group | Phase I: Pazopanib 200 mg /Lapatinib 1500 mg | Phase I: Pazopanib 800 mg /Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
grams per liter (g/L) | -4.25 (4.573) | -6.17 (5.707) | -3.80 (1.924) | -5.17 (3.545) | -13.66 (16.959) | -7.17 (4.215)

21. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, and Lactate Dehydrogenase
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Groups:
- Phase I: Pazopanib 200 mg/Lapatinib 1500 mg: Pazopanib 200 mg OD and Lapatinib 1500 mg OD
- Phase I: Pazopanib 800 mg/Lapatinib 1500 mg: Pazopanib 800 mg OD and Lapatinib 1500 mg OD
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
International Units per Liter (IU/L)
  Alkaline phosphatase | 9.8 (11.47) | 22.8 (39.55) | 31.2 (53.60) | 15.8 (22.66) | 22.0 (28.54) | 22.0 (47.15)
  Alanine aminotransferase | 36.8 (66.35) | 139.5 (204.81) | 47.0 (48.09) | 33.2 (25.25) | 4.8 (7.19) | 47.7 (56.43)
  Aspartate aminotransferase | 15.0 (31.72) | 49.3 (71.63) | 13.8 (15.71) | 8.8 (7.03) | 13.5 (16.20) | 19.3 (18.47)
  Lactate dehydrogenase | 148.0 (96.42) | 127.0 (144.60) | 46.0 (35.86) | 321.2 (534.42) | 124.7 (136.46) | 116.8 (59.26)

22. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Amylase and Lipase
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
Units per liter (U/L)
  Amylase | 24.3 (36.42) | 24.4 (17.04) | 27.3 (66.4) | 31.0 (38.96) | 44.4 (52.52) | 23.3 (39.38)
  Lipase | 147.0 (292.02) | 23.3 (44.98) | 33.0 (56.79) | 151.8 (230.63) | 67.3 (101.83) | 7.8 (21.09)

23. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Total Bilirubin and Creatinine
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/l)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
micromoles per liter (µmol/l)
  Total bilirubin | -0.000 (4.6307) | 2.613 (2.5162) | 3.368 (2.1520) | 6.130 (6.0799) | 4.135 (3.8089) | 6.398 (3.8952)
  Creatinine | 4.420 (15.3113) | 8.367 (11.3656) | 7.336 (6.6049) | 6.893 (6.6297) | 9.727 (9.7448) | 12.005 (19.3179)

24. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Calcium, Glucose, Potassium, Magnesium, Inorganic Phosphorus, Sodium, and Urea
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/l)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
millimoles per liter (mmol/l)
  Calcium | -0.062 (0.0250) | -0.045 (0.1173) | 0.036 (0.0572) | 0.061 (0.0874) | 0.047 (0.1155) | -0.014 (0.1166)
  Glucose | 0.56 (1.385) | 3.35 (6.653) | 1.20 (1.114) | 1.02 (2.654) | 1.55 (0.589) | 0.65 (0.934)
  Potassium | 0.075 (0.4992) | 0.400 (0.3033) | 0.420 (0.3033) | 0.500 (0.2608) | 0.600 (0.5967) | 0.183 (0.2229)
  Magnesium | 0.069 (0.0237) | -0.019 (0.0573) | 0.058 (0.0463) | 0.051 (0.0510) | 0.043 (0.0615) | 0.056 (0.0920)
  Sodium | -1.000 (1.8257) | 0.500 (2.0736) | 1.800 (1.6432) | 1.333 (2.0656) | 1.500 (4.5497) | 0.000 (0.6325)
  Urea | 1.9 (0.18) | 0.6 (1.18) | 0.8 (1.74) | 1.1 (1.27) | 0.9 (1.20) | 1.7 (1.72)
  Inorganic phosphorus | 0.02 (0.168) | 0.11 (0.186) | 0.41 (0.553) | 0.16 (0.164) | 0.01 (0.129) | 0.25 (0.185)

25. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Thyroxine
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/l)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
picomoles per liter (pmol/l) | -0.740 (2.8496) | -1.498 (1.8681) | 1.105 (3.6173) | 1.879 (2.8191) | 0.377 (3.9731) | -0.781 (1.0040)

26. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Free T3 (Triiodothyronine)
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: All-treated Population for Phase I. Data are presented for only those participants who provided chemistry measurements at both baseline and post-baseline. For some arms, data were not collected for either baseline or post-baseline assessments.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/l)
Arm/Group | Phase I: Pazopanib 200 mg /Lapatinib 1500 mg | Phase I: Pazopanib 800 mg /Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 0 | 0 | 5 | 0 | 6 | 0
picomoles per liter (pmol/l) |  |  | -0.07 (0.222) |  | -0.94 (1.291) |

27. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Thyroid Stimulating Hormone
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: milliunits per liter (mU/L)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
milliunits per liter (mU/L) | -0.5068 (1.99588) | 0.1900 (0.38931) | 0.6543 (0.73309) | 0.6660 (0.70497) | 0.6080 (11.10117) | 2.2940 (1.25335)

28. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Total T3
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/l)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 0 | 7 | 0 | 0
nanomoles per liter (nmol/l) | -0.071 (0.1113) | 0.214 (0.2851) |  | 0.004 (0.0028) |  |

29. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Hemoglobin
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: All-treated Population for Phase I. Data are presented for only those participants who provided hematology measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 6 | 6
grams per Liter (g/L) | -7.25 (14.975) | -7.83 (12.999) | -4.80 (9.834) | -3.33 (13.095) | -16.17 (9.867) | -21.02 (59.642)

30. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Hematocrit
Description: as for outcome 16
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 6 | 6
percent | -0.02 (0.034) | -0.02 (0.029) | -0.02 (0.023) | 0.00 (0.027) | -0.09 (0.103) | 0.01 (0.024)

31. Primary Outcome: Mean Change From Baseline to Maximum Value in the Study for Lymphocytes, Neutrophils, Platelet Count, and White Blood Count
Description: Change from baseline is calculated as the maximum changed value in the study minus the value at Baseline.
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: giga (10^9) per liter (GI/L)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 6 | 6
giga (10^9) per liter (GI/L)
  Lymphocytes, n=3, 6, 4, 6, 6, 6 | -0.377 (0.4611) | -0.120 (0.4291) | -0.153 (0.3083) | -0.032 (0.2807) | -0.218 (0.2316) | -0.250 (0.3017)
  Total Neutrophils, n=3, 6, 4, 6, 6, 6 | -0.693 (1.0775) | -3.000 (3.2727) | -1.370 (1.5036) | -0.595 (0.8783) | -1.723 (1.7320) | -0.617 (2.7154)
  Platelet count, n=4, 6, 5, 6, 6, 6 | -12.3 (30.08) | -74.7 (74.18) | -65.4 (32.65) | -25.3 (40.00) | -35.5 (54.72) | -61.8 (32.17)
  White blood cell count, n=4, 6, 5, 6, 6, 6 | -0.845 (1.0849) | -2.933 (3.6335) | -1.950 (2.1249) | -0.850 (0.9072) | -1.717 (2.2355) | -0.850 (2.4468)

32. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for International Normalized Ratio (Prothrombin Time)
Description: as for outcome 18
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: All-treated Population for Phases I and II. Data are presented for only those participants who provided hematology measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 6 | 5
ratio | 0.077 (0.0866) | -0.023 (0.0638) | 0.056 (0.0472) | 0.000 (0.1097) | 0.015 (0.0764) | 0.006 (0.0134)

33. Primary Outcome: Mean Change From Baseline to Maximum Value in Phase I of the Study for Partial Thromboplastin Time and Prothrombin Time
Description: as for outcome 19
Time Frame: Baseline to study completion (up to 844 days for Phase I)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 6 | 5
seconds (sec)
  Partial thromboplastin time | 1.10 (1.299) | 2.88 (1.986) | 2.62 (5.545) | -0.38 (6.122) | 2.18 (2.082) | 1.00 (1.093)
  Prothrombin time | 0.38 (0.532) | 0.47 (0.940) | 0.64 (0.981) | -0.02 (0.796) | 1.07 (1.722) | 0.56 (0.885)

34. Primary Outcome: Number of Participants Experiencing a Dose-limiting Toxicity at the Indicated Dose
Description: A dose-limiting toxicity (DLT) is defined as predefined adverse events or events that prevented participants from receiving 75% of their scheduled doses or from starting their next treatment period. The dose at which no more than 1 out of 6 participants experiences a DLT is defined as the optimally tolerated regimen. The OTR is important because it determines the highest dose combination that can be given without significant toxicity.
Time Frame: Cycle 1 in Phase I (up to Day 28)
Population: All-treated Population for Phase I
Measure: Number; unit: participants
Arm/Group | Phase I: Pazopanib 200 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 1500 mg | Phase I: Pazopanib 800 mg/Lapatinib 500 mg | Phase I: Pazopanib 800 mg/Lapatinib 750 mg | Phase I: Pazopanib 800 mg/Lapatinib 1000 mg | Phase I: Pazopanib 600 mg/Lapatinib 1000 mg
Number analyzed (Participants) | 4 | 6 | 5 | 7 | 6 | 6
participants | 0 | 1 | 1 | 1 | 1 | 1

35. Primary Outcome: Overall Response (OR) in Phase II Based GlaxoSmithKline's Evaluation
Description: OR is the number of participants whose response was classified as a complete response or partial response (disappearance of enhancing tumor (ET) or reduction of ET by >=50%, respectively, on consecutive scans [CS] >=1 month (m) apart, off steroids, and neurologically stable/improved), progressive disease (increase of ET of >=25% on CS >=1 m apart or neurologically worse, and steroids stable/increased), or stable disease (all other situations) per MacDonald criteria. Participants were evaluated with magnetic resonance imaging. Baseline and the 4- and 8-w assessments are categorized as <8 w.
Time Frame: Date of first dose of study drug to date of documented and confirmed progression, or to date of death due to any cause (assessed at baseline, 4 and 8 weeks, and every 8 weeks thereafter until study withdrawal; up to Day 878)
Population: All-treated Population in Phase II who also had a response assessment
Measure: Number; unit: participants
Groups:
- Phase II: Biomarker Positive: All participants received pazopanib 400 mg twice daily (BID) and lapatinib 1000 mg OD. Biomarker-positive participants were those who expressed EGFRvIII and/or PTEN.
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
participants
  Complete response | 0 | 0
  Partial response | 1 | 2
  Stable disease, >=8 weeks | 7 | 6
  Progressive disease, <8 weeks | 7 | 8
  Progressive disease | 4 | 6

36. Primary Outcome: Overall Response (OR) in Phase II Based on the Investigator-assigned Response
Description: as for outcome 35
Time Frame: as for outcome 35
Population: All-treated Population for Phase II who also had a response assessment.
Measure: Number; unit: participants
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
participants
  Complete response | 0 | 0
  Partial response | 1 | 1
  Stable disease, >=8 weeks | 7 | 7
  Progressive disease, <8 weeks | 7 | 9
  Progressive disease | 4 | 5

37. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) analysis was performed on all participants. PFS is presented as the number of participants experiencing disease progression or death due to any cause. Participants who are alive and have not progressed at the time of analysis are considered censored, and the date associated with the last visit with disease assessment will be used.
Time Frame: Date of the first dose of study drug to the date of documented and confirmed progression by Mac Donald criteria, or to date of death due to any cause (up to Day 878)
Population: All-treated Population for Phase II
Measure: Number; unit: participants
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
participants
  Disease progression | 15 | 18
  Death | 0 | 2
  Censored | 4 | 2

38. Secondary Outcome: Time to Disease Progression or Death Due to Any Cause
Time Frame: as for outcome 37
Population: All-treated Population for Phase II
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
days | 62 [56 to 90] | 56 [45 to 113]

39. Primary Outcome: Overall Response (OR) in Phase II Based on an Independent Radiologist's Review
Description: as for outcome 35
Time Frame: as for outcome 35
Population: All-treated Population for Phase II who also had a response assessment
Measure: Number; unit: participants
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
participants
  Complete response | 0 | 0
  Partial response | 0 | 0
  Stable disease, >=8 weeks | 5 | 4
  Progressive disease, <8 weeks | 5 | 8
  Progressive disease | 4 | 6
  Unconfirmed partial response | 4 | 4

40. Primary Outcome: Progression-free Survival at 6 Months
Description: Progression-free survival (PFS) analysis was performed on all participants. PFS is presented as the number of participants experiencing disease progression or death due to any cause. Participants who are alive and have not progressed at the time of analysis are considered censored, and the date associated with the last visit with disease assessment will be used. The participants who are still alive and whose follow-up extends to at least 6 months are considered At Risk.
Time Frame: Date of the first dose of study drug to 6 months
Population: All-treated Population for Phase II
Measure: Number; unit: participants
Arm/Group | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Number analyzed (Participants) | 19 | 22
participants
  Disease progression at or prior to 6 months | 15 | 16
  Death at or prior to 6 months | 0 | 2
  Censored at or prior to 6 months | 4 | 1
  At risk beyond 6 months | 0 | 3

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AES in Phases I and II were collected from Day 1 of study treatment to study completion (up to 844 days for Phase I; up to 878 days for Phase II).
Groups:
- Phase II: Biomarker Positive: All participants received pazopanib 400 mg twice daily (QD) and lapatinib 1000 mg QD. Biomarker-positive participants were those who expressed epithelial growth factor receptor vIII (EGFRvIII) and/or phosphate and tensin homolog (PTEN).
- Phase II: Biomarker Negative: All participants received pazopanib 400 mg QD and lapatinib 1000 mg QD. Biomarker-negative participants were those who did not express either EGFRvIII and/or PTEN.
Arm/Group | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg | Phase II: Biomarker Positive | Phase II: Biomarker Negative
Serious Adverse Events (participants affected / at risk) | 15/34 | 6/19 | 8/22
Other Adverse Events (participants affected / at risk) | 33/34 | 18/19 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg (N=34) | Phase II: Biomarker Positive (N=19) | Phase II: Biomarker Negative (N=22)
Convulsion (Nervous system disorders) | 1 | 1 | 4
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Cerebral hemorrhage (Nervous system disorders) | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Pazopanib 200-800 mg/Lapatinib 500-1500 mg (N=34) | Phase II: Biomarker Positive (N=19) | Phase II: Biomarker Negative (N=22)
Diarrhea (Gastrointestinal disorders) | 19 | 12 | 14
Fatigue (General disorders) | 16 | 11 | 10
Headache (Nervous system disorders) | 9 | 7 | 8
Hypertension (Vascular disorders) | 9 | 3 | 9
Nausea (Gastrointestinal disorders) | 9 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 8 | 4
Vision blurred (Eye disorders) | 9 | 1 | 5
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5 | 6
Convulsion (Nervous system disorders) | 4 | 2 | 4
Alanine aminotransferase increased (Investigations) | 8 | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 6
Confusional state (Psychiatric disorders) | 0 | 4 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3
Constipation (Gastrointestinal disorders) | 4 | 1 | 4
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 4
Lipase increased (Investigations) | 3 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Somnolence (Nervous system disorders) | 2 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4
Blood amylase increased (Investigations) | 1 | 3 | 2
Hyperbilirubinaemia/blood bilirubin increased (Hepatobiliary disorders) | 1 | 1 | 5
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 3
Speech disorder (Nervous system disorders) | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 3
Mood altered/mood swings (Psychiatric disorders) | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 4 | 3 | 3
Amnesia (Nervous system disorders) | 4 | 5 | 1
Aphasia (Nervous system disorders) | 4 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 2
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 2 | 2
Cushingoid (Endocrine disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 1
Mucosal inflammation (General disorders) | 3 | 1 | 1
Edema peripheral (General disorders) | 3 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 1 | 5
Decreased appetitie (Metabolism and nutrition disorders) | 3 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 2 | 3 | 4
Peripheral motor neuropathy (Nervous system disorders) | 2 | 3 | 3
Pyramidal tract syndrome (Nervous system disorders) | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 2 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2
Ataxia (Nervous system disorders) | 1 | 2 | 4
Cranial nerve disorder (Nervous system disorders) | 1 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 2 | 1
Hemiparesis (Nervous system disorders) | 3 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 2
Partial seizures (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hair color changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Blood urea increased (Investigations) | 1 | 0 | 3
Weight decreased (Investigations) | 1 | 2 | 1
Weight increased (Investigations) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Candidiasis (Infections and infestations) | 1 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.